CLINICAL TRIAL: NCT03514316
Title: Scalpel Versus Laser Gingivectomy in the Management of Periodontal Health During Orthodontic Treatment: a Randomized Controlled Clinical Trial
Brief Title: Scalpel Versus Laser Gingivectomy in Orthodontic Patients in the Management of Periodontal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Andrea Noviello, Post graduate Student, Department of Orthodontics, Department of Clinical Sciences and Translational Medicine, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206/17
Record Dates: First submitted 2018-04-11; First posted 2018-05-02 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Orthodontic Appliance Complication; Gingival Overgrowth
Keywords: gingival overgrowth; diode laser gingivectomy; scalpel gingivectomy; orthodontic treatment
MeSH Terms: conditions — Gingival Overgrowth

STUDY DESIGN:
Intervention Model Description: a prospective three-arm parallel group randomized clinical trial with 1:1:1 allocation ratio
Who Masked: Outcomes Assessor
Masking Description: The observer who performed all the measurements was blinded to the group assignment. The study was blinded in regard to the statistical analysis: blinding was obtained by eliminating from the elaboration file every reference to patient group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scalpel Gingivectomy (Active Comparator): Patients treated with Scalpel Gingivectomy on the labial side of the anterior maxillary teeth
  Interventions: Procedure: Scalpel Gingivectomy
- Laser Gingivectomy (Active Comparator): Patients treated with Laser Gingivectomy on the labial side of the anterior maxillary teeth
  Interventions: Procedure: Laser Gingivectomy
- Nonsurgical periodontal treatment (Active Comparator): Patients treated with a full-mouth periodontal debridement
  Interventions: Procedure: Nonsurgical periodontal treatment

INTERVENTIONS:
Procedure: Scalpel Gingivectomy — The patients were anesthetized in the area around the teeth which were to undergo the procedure with local anesthesia (Drug: 2% lidocaine and 1:80,000 adrenaline). Initially, the Periodontal Probing Depth was measured and when sufficient anesthesia was achieved, biologic width calculation was done by the trans-gingival probing method. Once the amount of gingival tissue to be excised was demarcated, an external bevel incision was performed by using a scalpel blade (Device: scalpel blade No.15) and the gingival tissue was excised. Left out tissue tags and any beads of granulations tissue were removed to attain a smooth surface.
  Arms: Scalpel Gingivectomy
Procedure: Laser Gingivectomy — In the Laser Gingivectomy group, the procedure was performed by using a 810 nm diode laser (Device: 810 nm FOX III diode laser) . Though a local anesthetic gel is sufficient considering that the procedure is minimally invasive, the area was adequately anesthetized with 2% lidocaine and 1:80,000 adrenaline. The laser unit, comprising of a 300 μm disposable tip, was used in a contact mode with a setting of 1 to 1.5 watts in continuous mode along the demarcated area with a paint brush like strokes progressing slowly to remove the gingival tissue and expose adequate amount of tooth structure. High-volume suction was used to evacuate the laser plume and charred odor
  Arms: Laser Gingivectomy
Procedure: Nonsurgical periodontal treatment — In all subjects of the Control Group a full-mouth periodontal debridement was performed at baseline, 1 and 3 months with an ultrasonic scaler. Chlorhexidine prophylaxis (0.05% chlorhexidine gluconate) was also administered twice a day for 2 weeks after the periodontal treatment. Oral-hygiene instructions were reinforced again.
  Arms: Nonsurgical periodontal treatment

SUMMARY:
Patients undergoing orthodontic treatment with fixed appliances usually develop gingival enlargement (GE). Its development is usually attribute to chronic inflammation, and may cause both esthetic and functional problems for the patient. In many cases, the gingival hyperplasia demands periodontal surgery in order to increase the length of the crown during or after the orthodontic treatment. Previously conventional surgical procedures were performed using a scalpel under local anaesthesia for these procedures. Lately the use of laser has been proposed. The majority of the studies comparing laser gingivectomy with scalpel gingivectomy show some limits: they are not randomized, they are not prospective, and they have no control group. The primary objective of the present investigation was to conduct a randomized controlled trial (RCT) evaluating the effectiveness of diode laser gingivectomy versus scalpel gingivectomy in the management of periodontal health among patients receiving fixed orthodontic appliance therapy, compared with a non surgical control group.

DETAILED DESCRIPTION:
Gingival enlargement (GE) is one of the most common soft tissue problems in patients undergoing orthodontic fixed treatment, particularly when spaces are rapidly closed and oral hygiene is poor. The mechanism by which GE occurs during orthodontic treatment is not fully understood. The initiation and development of periodontal disease depend on a dynamic equilibrium between the microbial challenge and the host's immune-inflammatory responses. The presence of fixed appliances influences plaque accumulation around the retentive components attached to the teeth and the colonization of important periodontopathic bacteria. Chronic inflammation of the soft tissues is caused by a significant increase in edema and inflammatory cells that can influence the sub-gingival ecosystem by creating an appropriate anaerobic environment, leading to a shift in the composition of the microflora. When gingival tissues are enlarged, varying from mild enlargement of isolated interdental papillae to segmental or uniform and marked enlargement affecting one or both jaws, the tooth surfaces become difficult to access, inhibiting good oral hygiene and resulting in more inflammation and bleeding because enlarged gingival tissues. In artificially deeper periodontal pockets, the root surfaces are contaminated with an accumulation of plaque and calculus, as well as infiltration of bacteria and bacterial endotoxins into cementum. Complete removal of these harmful substances is essential for the healing of periodontal tissue. However, nonsurgical periodontal treatment (including oral hygiene instruction, scaling, root planing, and prophylaxis) is not always effective when GE is extensive and self-care is compromised. When GE further impedes the maintenance of oral hygiene (thereby resulting in further damage to periodontal tissues), causes aesthetic and functional problems, and compromises orthodontic tooth movement, it is necessary to provide additional surgery treatment such as gingivectomy, in order to correct gingival border contours. Gingivectomy can be performed by conventional scalpels, electrosurgery, chemosurgery, and laser. Preservation of biologic width is the therapeutic endpoint of all these procedures. 3 mm of tooth structure above the osseous crest is considered safe to prevent any attachment loss. The conventional surgery performed by a small scalpel has been considered the most common method because of its ease of use, accuracy, and minimal damage to tissues. However, scalpels do not provide a good hemostasis, which is important on highly perfused tissues such as in the oral cavity. The advent of diode lasers highly absorbable by melanin and hemoglobin allows soft-tissue manipulations providing sound results in periodontal surgery, tissue alterations related to orthodontic treatment, and oral lesions. The diode laser separates and coagulates at the same time, facilitating immediate hemostasis and resulting in minimal bleeding. Healing is rapid and there is reduced potential for infection. The diode laser has an affinity for only soft tissue, thereby preventing damage to the surrounding bone and enamel. Therefore, using diode lasers might be advantageous because of better control, potentially lower pain and inflammation, and improved wound healing. In literature, no studies directly compared conventional scalpel surgery versus diode laser-assisted surgery in orthodontic patients with GE. Moreover, the majority of the studies comparing laser gingivectomy with scalpel gingivectomy show some limits: they are not randomized, they are not prospective, and they have no control group. Therefore, the aim of the present study was to compare the use of the 810nm diode laser with conventional surgery and to evaluate the effectiveness of gingivectomy as an adjunct to nonsurgical periodontal treatment in the management of GE during orthodontic treatment. The Consolidated Standards of Reporting Trials (CONSORT) checklist was used as a guideline for conducting and reporting this trial. The present Randomized Clinical Trial was designed as a prospective three-arm parallel group randomized clinical trial with 1:1:1 allocation ratio. The study was approved by the Ethics Committee at the University of Rome "Tor Vergata", (protocol number 206/17), and informed consent was obtained from the patients' parents. A total of 60 (33 Males; 27 Females) subjects, with a mean age of 14.4 ± 1.9 years (range 11.7-19.8 years), undergoing orthodontic treatment at the Department of Orthodontic of the University of Rome "Tor Vergata" were recruited for the study. Gingival overgrowth diagnosis was defined as presence of quadratic anterior teeth (crown width/length ratio ≤0.85), gingival margin located incisal to the tooth cervical convexity and presence of mean Probing Pocket Depths (PPD) ≥ 4mm coronal to the cement-enamel junction (CEJ) at three buccal points around each tooth of the anterior segment (mesial, mid-point, distal). Crown Width (CW) and Clinical Crown Length (CCL) were measured pre-operatively with a digital caliper: CCL, measured as the distance between incisal edge and gingival margin along the tooth long axis; CW measured at the point between incisal and middle third of CCL. All subjects received ongoing nonsurgical periodontal treatment and instructions on oral hygiene. After the conventional management approach for gingival enlargement, patients with persistent gingival overgrowth were enrolled in the study and blindly assigned to three groups. In the first group (TG1), all subjects underwent a conventional scalpel gingivectomy of the maxillary anterior sextant. In the second group (TG2), all subjects were treated using laser-assisted gingivectomy; while subjects assigned to the third group underwent only nonsurgical periodontal treatment and served as the control group (CG). Both TGs were consecutively treated by one clinician. The PPDs were recorded to determine the biologic width and to assess how much tissue could be contoured without involving osseous surgery, using a North Carolina periodontal probe. Remembering that there exists a 3.0 mm biologic zone, the maximum amount of tissue removal could be calculated. The periodontal probe was placed apically to the alveolar crest, and the marginal gingival level was measured. An explorer was used to mark reference spots of the biologic zone, serving as the visual finishing point. At baseline (before surgery) all patients of the three groups underwent a full periodontal screening. Their oral hygiene and gingival inflammation were assessed using CCL, PPD, Plaque Index (PI) and Gingival Index (GI) at three buccal points around each tooth of the anterior segment (mesial, mid-point, distal). All measures were repeated at 1, 3 and 6 months post-surgery or nonsurgical periodontal treatment. Overall patient data were calculated as mean value by averaging measurements in all sites of six upper anterior teeth. A sample size for this trial was calculated according to the method proposed by Whitehead et al. For a standardized effect size of 1 (a clinically relevant change of 0.75 mm with a combined SD of 0.68 mm derived from Mavroggianis et al.) for the primary outcome variable PPD at 3 months, a sample size of 17 subjects per group was required for a type I error rate of 5% and a power of 80%. To account for potential dropouts, 20 subjects per group were recruited. Allocation of patients to the three groups was determined by a computer-generated randomization list using Rv.0.1 software and by a block size of 4. Then, the allocation information (randomization results) was concealed in opaque and sealed envelopes by the statistician. The observer who performed all the measurements was blinded to the group assignment. The study was blinded in regard to the statistical analysis: blinding was obtained by eliminating from the elaboration file every reference to patient group assignment. Reliability of the periodontal assessments was conducted among 10 patients throughout the study. Exploratory statistics revealed that all periodontal variables were normally distributed (Kolmogorov-Smirnov test) with equality of variances (Levene's test). All statistical computations were performed with SPSS software (Statistical Package for the Social Sciences, SPSS, Version 12, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* overgrown gingivae on the labial side of the anterior teeth secondary to fixed appliance therapy,
* six maxillary anterior teeth present,
* healthy nonsmokers patients.

Exclusion Criteria:

* patients with poor oral hygiene;
* patients with mucogingival infection;
* patients taking medications that may cause drug-associated gingival enlargement (eg. calcium channel blockers, anticonvulsants, or immunosuppressants)
* patients currently pregnant or lactating;
* patients with any medical condition affecting wound healing.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth Changes after Scalpel Gingivectomy vs Laser Gingivectomy compared with a Control Group receiving non surgical periodontal treatment only at 3 time points respect to baseline. | 6 months
  The primary outcome is the reduction of the Pocket Depth. The objective is to evaluate the change in the Pocket Depth induced by Scalpel Gingivectomy or Laser Gingivectomy, compared with a nonsurgical periodontal treatment group at 3 time points respect to baseline: 1 month, 3 months and 6 months.
  Probing Pocket Depths (PPDs) were recorded at baseline to determine the biologic width and to assess how much tissue could be contoured without involving osseous surgery, using a North Carolina periodontal probe; Scalpel Gingivectomy or Laser Gingivectomy were performed in the treated groups.
  In the non surgical periodontal treatment group, full-mouth periodontal debridement was performed at baseline, 1 and 3 months with an ultrasonic scaler.
  Overall patient data were calculated as mean value by averaging measurements in all sites of six upper anterior teeth.

SECONDARY OUTCOMES:
Increased Clinical Crown Length (CCL) after Scalpel Gingivectomy vs Laser Gingivectomy | 6 months
  The secondary outcome is the increase of the CCL, measured as the distance between incisal edge and gingival margin along the tooth long axis.
  The objective is to evaluate the change in the CCL induced by Scalpel Gingivectomy or Laser Gingivectomy, compared with a nonsurgical periodontal treatment group.
  All measures were repeated at 1, 3 and 6 months post-surgery or full-mouth periodontal debridement. Overall patient data were calculated as mean value by averaging measurements of six upper anterior teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Noviello, Principal Investigator — Department of Orthodontics, Department of Clinical Sciences and Translational Medicine, University of Rome "Tor Vergata," Rome, Italy
Locations (1):
- Department of Orthodontics, Department of Clinical Sciences and Translational Medicine, University of Rome "Tor Vergata"., Roma, Italy

REFERENCES:
- [Background] To TN, Rabie AB, Wong RW, McGrath CP. The adjunct effectiveness of diode laser gingivectomy in maintaining periodontal health during orthodontic treatment. Angle Orthod. 2013 Jan;83(1):43-7. doi: 10.2319/012612-66.1. Epub 2012 May 16. PMID 22591260
- [Background] Silva CO, Soumaille JM, Marson FC, Progiante PS, Tatakis DN. Aesthetic crown lengthening: periodontal and patient-centred outcomes. J Clin Periodontol. 2015 Dec;42(12):1126-34. doi: 10.1111/jcpe.12482. Epub 2015 Dec 23. PMID 26613260
- [Background] Mavrogiannis M, Ellis JS, Seymour RA, Thomason JM. The efficacy of three different surgical techniques in the management of drug-induced gingival overgrowth. J Clin Periodontol. 2006 Sep;33(9):677-82. doi: 10.1111/j.1600-051X.2006.00968.x. Epub 2006 Jul 20. PMID 16856895
- [Background] Farista S, Kalakonda B, Koppolu P, Baroudi K, Elkhatat E, Dhaifullah E. Comparing Laser and Scalpel for Soft Tissue Crown Lengthening: A Clinical Study. Glob J Health Sci. 2016 Oct 1;8(10):55795. doi: 10.5539/gjhs.v8n10p73. PMID 27302447
- [Background] Volchansky A, Cleaton-Jones P. Clinical crown height (length)--a review of published measurements. J Clin Periodontol. 2001 Dec;28(12):1085-90. doi: 10.1034/j.1600-051x.2001.281201.x. PMID 11737504
- [Background] Mavrogiannis M, Ellis JS, Thomason JM, Seymour RA. The management of drug-induced gingival overgrowth. J Clin Periodontol. 2006 Jun;33(6):434-9. doi: 10.1111/j.1600-051X.2006.00930.x. PMID 16677333
- [Background] McGuire MK, Scheyer ET. Laser-assisted flapless crown lengthening: a case series. Int J Periodontics Restorative Dent. 2011 Jul-Aug;31(4):357-64. PMID 21837301
- [Background] Ize-Iyamu IN, Saheeb BD, Edetanlen BE. Comparing the 810nm diode laser with conventional surgery in orthodontic soft tissue procedures. Ghana Med J. 2013 Sep;47(3):107-11. PMID 24391225
- [Background] Gong Y, Lu J, Ding X. Clinical, microbiologic, and immunologic factors of orthodontic treatment-induced gingival enlargement. Am J Orthod Dentofacial Orthop. 2011 Jul;140(1):58-64. doi: 10.1016/j.ajodo.2010.02.033. PMID 21724088
- [Background] Zanatta FB, Ardenghi TM, Antoniazzi RP, Pinto TM, Rosing CK. Association between gingivitis and anterior gingival enlargement in subjects undergoing fixed orthodontic treatment. Dental Press J Orthod. 2014 May-Jun;19(3):59-66. doi: 10.1590/2176-9451.19.3.059-066.oar. PMID 25162567
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Derived] Lione R, Pavoni C, Noviello A, Clementini M, Danesi C, Cozza P. Conventional versus laser gingivectomy in the management of gingival enlargement during orthodontic treatment: a randomized controlled trial. Eur J Orthod. 2020 Jan 27;42(1):78-85. doi: 10.1093/ejo/cjz032. PMID 31111882